CLINICAL TRIAL: NCT05264649
Title: Effect of Acupuncture vs Chinese Medicine vs Combined Therapy on Aromatase Inhibitor-related Arthralgia Among Women With Early-Stage Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lee I-Ting, doctor, Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1100903
Record Dates: First submitted 2022-02-20; First posted 2022-03-03 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Arthralgia
Keywords: aromatase inhibitors-associated arthralgia; aromatase inhibitors; breast cancer; musculoskeletal disorders; hormonal anti-estrogen therapy; endocrine therapy
MeSH Terms: conditions — Arthralgia; Breast Neoplasms; Musculoskeletal Diseases | interventions — Acupuncture Therapy; guizhi-shaoyao-zhimu decoction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acupuncture group (Experimental): Stainless steel, disposable, sterile needles choosing based on the needs of different body parts (0.22 gauge x 25mm, 0.22 gauge x 40mm, or 0.25 gauge x 100mm) were inserted to acupoints at traditional depths and angles.
  Interventions: Device: acupuncture
- Chinese medicine group (Experimental): The Chinese medicine group used Guizhi-Shaoyao-Zhimu decoction (GZSD) as their medical intervention. The GZSD samples were made and packed by Sun Ten Pharmaceutical Co. Ltd., a firm that meets the requirements of the good manufacturing practice (GMP) certification in Taiwan. Every 4g of concentrated GZSD was sealed in an isolated paper drug bag.
  Interventions: Drug: Guizhi-Shaoyao-Zhimu decoction
- combined group (Experimental): The combined group would have both acupuncture and Chinese medicine interventions.
  Interventions: Device: acupuncture; Drug: Guizhi-Shaoyao-Zhimu decoction

INTERVENTIONS:
Device: acupuncture — The acupuncture group were consisted of twelve 30 minutes sessions 2 times per week sessions for 6 weeks. The acupoints were included full body protocol (LI4, LR3, and PC7) and joint-specific protocol tailored as many as three of the patient's most painful joint areas. After 20 minutes "De Qi" reported by patients, needles were restimulated manually and removed after an additional 10 minutes.
  Arms: acupuncture group; combined group
Drug: Guizhi-Shaoyao-Zhimu decoction — The patients consumed GZSD (4g paper bagged medicine) three times per day (total daily dose was 12 g/day) continuously during the 6-week intervention period.
  Arms: Chinese medicine group; combined group

SUMMARY:
Aromatase inhibitors have been used to treat hormone receptor positive breast cancer women in menopause, but side effects, such as joint pain, would affect their qualities of life. Chinese herbs or acupuncture provides promising clinical effects and plays an important role on alleviating the side effects of cancer treatment. This clinical trial will evaluate the effect of the acupuncture, Chinese medicine, and the combination of both on joint pain related to aromatase inhibitors among women with early-stage breast cancers.

DETAILED DESCRIPTION:
Reduce estrogen exposure can lower the risk of breast cancer recurrence. Aromatase inhibitors have been used to treat hormone receptor positive breast cancer women in menopause for years. It can increase the survival rate and decrease the chance of recurrence. However, many patients suffered from the side effects of medication, including joint pain, is the main reason for decreasing medication adherence and influencing patients' quality of life. Based on previous phase III clinical trial study, acupuncture may relieve aromatase inhibitor associated joint pain, and experts believe that acupuncture could also be considered as an effective adjuvant treatment. Chinese herbs or acupuncture provides promising clinical effects and plays an important role in alleviating the side effects of cancer treatment. Guizhi-Shaoyao-Zhimu decoction has frequently being prescribed to treat joint pain in traditional Chinese medicine practice. The design of this clinical trial will evaluate the effects of the acupuncture, Chinese medicine, and the combination of both on joint pain related to aromatase inhibitors among women with early-stage breast cancer. The goal of this study was to evaluate the efficacy and safety with regards to utilizing acupuncture and Chinese herbs in treating joint pain related to the usage of aromatase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Women with diagnosis of early breast cancer (stages I-III), expressing hormone receptor-positive (ER+, PR+, or both) and took third generation aromatase inhibitors (AIs).
2. Post- or pre-menopausal with the use of a gonadotropin-releasing hormone agonist.
3. Taking AIs for more than 30 days before registration and planned to continue treatment for over 1 year.
4. Have already been recovered from the surgery or chemotherapy.
5. Have a ECOG performance status score of 0 to 1.
6. Joint pain which has developed or worsened since starting AIs therapy. The worst pain item score of Brief Pain Inventory-Short Form (BPI-SF) is at least 3 and above.
7. Have a Eastern Cooperative Oncology Group (ECOG) grading scale for chemotherapy-induced peripheral neuropathy score of 1 to 2.
8. The patient could cooperate the intervention and sign the informed consent.

Exclusion Criteria:

1. Had received acupuncture treatment for joint pain would be excluded, but patients with acupuncture treatment for less than 2 times due to other reasons could be included.
2. Had a history of fractures or underwent surgery on the knee or hand joints in the past six months.
3. Had severe bleeding disorders. The platelet counts are below 50,000 per μl.
4. Cognitive disorders (included dementia).
5. Lymphedema after breast cancer surgery.

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2023-03-03 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory-Worst Pain Item (BFI-WP) | Change from baseline at 6 weeks
  a 0- to 10-point scale (0 [no pain] to 10 [pain as bad as you can imagine)

SECONDARY OUTCOMES:
Brief Pain Inventory - Short Form (BPI-SF) | Change from baseline at 6 weeks
  The Brief Pain Inventory-Short Form (BPI-SF) was used to evaluate the worst pain, pain severity, and pain- related interference scores. (0 [no pain] to 10 [pain as bad as you can imagine)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from baseline at 6 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was used in the evaluation of pain (score range, 0-20), stiffness (score range, 0-8), physical function of lower limb (score range, 0-68).
Modified Score for the Assessment and Quantification of Chronic Rheumatoid Affections of the Hands (M-SACRAH) | Change from baseline at 6 weeks
  Affections of the Hands (M-SACRAH) was used in the evaluation of pain, stiffness, physical function of upper limb.
Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) | Change from baseline at 6 weeks
  The Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) measured physical and functional well- being and endocrine symptoms (score range, 0-128)

CONTACTS AND LOCATIONS:
Overall Officials: I-Ting Lee, Bachelor, Principal Investigator — Show Chwan Memorial Hospital
Locations (1):
- ShowChwanMH, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided